CLINICAL TRIAL: NCT04535050
Title: A Prospective, Multicenter, Sham-controlled, Single-blinded, Randomized, Pilot Study to Evaluate the Safety and Effectiveness of DENEX Renal Denervation System in Patients With Uncontrolled Hypertension Not Treated With Anti-HTN Medication
Brief Title: DENEX Renal Denervation in Patients With Hypertension on no Antihypertensive Medications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kalos Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DN_E101
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Renal Denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DENEX Renal denervation (Experimental): Subjects are treated with the renal denervation procedure after randomization
  Interventions: Device: Renal denervation
- Sham control (Sham Comparator): Subjects are treated with renal angiography
  Interventions: Procedure: Renal angiography

INTERVENTIONS:
Device: Renal denervation — Renal Denervation: DENEX system
  Arms: DENEX Renal denervation
Procedure: Renal angiography — Renal angiography
  Arms: Sham control

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of renal denervation using DENEX System in patients with hypertension without antihypertensive medication, compared with the sham group.

DETAILED DESCRIPTION:
DENEX system developed by Kalos Medical Inc. is a renal denervation system to efficiently block the sympathetic nerve of the kidney with minimal invasive procedure. It was developed to block the sympathetic nerves distributed in blood vessel wall by delivering high frequency energy to the renal artery for the purpose of treating hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 18 to 80 years old at the time of signing the informed consent
2. Subject who is drug-naïve or willing to discontinue current antihypertensive treatment (not on antihypertensive medications for at least 4 weeks prior to Screening Visit 1) at Screening Visit 1 through the 3-month post-procedure visit. Drug-naïve is defined as those with no previous exposure to antihypertensive medications.
3. Subject who meets all of the following blood pressure measurements:

   * Office Systolic Blood Pressrue (SBP) < 180 mmHg at Screening Visit 1
   * Office SBP ≥ 150 mmHg and < 180 mmHg, and office diastolic blood pressure (DBP) ≥ 90 mmHg at Screening Visit 2
   * 24-h ambulatory SBP ≥ 140 mmHg and < 170 mmHg at Screening Visit 2
4. Subject who voluntarily decides to participate in this clinical study and sign the written consent.
5. Subject who willing and able to complete all clinical investigation-related procedures and assessments

Exclusion Criteria:

1. Subject with renal anatomy that is ineligible for treatment:

   * Diameter of main renal artery for each kidney is < 3 mm or > 8 mm OR presence of accessory renal arteries (ARAs) with a diameter < 3 mm
   * Presence of fibromuscular dysplasia
   * Presence of kidney tumors or secretory tumors in the adrenal gland
   * > 50% stenosis in any treatable vessel
   * Presence of aneurysm (any localized increase in vessel diameter)
   * Treatment area within 5 mm segment in the renal artery contains an atheroma, calcification, or a renal artery stent
   * A single functioning kidney
   * Polycystic kidney disease
2. Subject with prior renal denervation, renal artery stenting, renal artery angioplasty, renal nephrectomy, or renal transplant
3. Subject with type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (HbA1c over 10.0%)
4. Subject with epidermal growth factor receptor (eGFR) < 45 mL/min/1.73 m2, using the 4-variable modification of diet in renal disease (MDRD) clinical investigation calculation
5. Subject taking sodium glucose co-transporter 2 (SGLT2) inhibitors or glucagon like peptide-1 (GLP-1) agonists that have been prescribed < 90 days prior to Screening Visit 1 or necessary to remain on these medications for duration of clinical investigation
6. Subject with ≥ 1 episode of orthostatic hypotension not related to medication changes within the past year prior to Screening Visit 1
7. Documented repeated (> 1) hospitalization for hypertensive crisis within the 12 months and/or any hospitalization for hypertensive crisis within the 3months prior to Screening Visit 1.
8. Subject requiring chronic oxygen support or mechanical ventilation (other than nocturnal respiratory support for sleep apnea)
9. Subject with primary pulmonary hypertension
10. Subject with untreated secondary cause of hypertension (known or suspected) or taking medications that increase sympathetic tone that could contribute to hypertension
11. Subject with frequent or chronic pain that requires treatment with NSAIDs for two or more days per week during the last month prior to Screening Visit 2 (aspirin and clopidogrel permitted for cardiovascular risk reduction)
12. Human immunodeficiency virus (HIV) on anti-retroviral drug therapy but without documentation that hypertension preceded initiation of anti-retroviral drug therapy
13. Subject with a history of myocardial infarction, stable or unstable angina, transient ischemic attack, cerebrovascular accident, heart failure, or atrial fibrillation within 3 months prior to Screening Visit 1
14. Subject who requires more than occasional use (e.g., PRN) of narcotic drugs over the month prior to Screening Visit 1
15. Subject currently taking anti-mineralocorticoid medications, unless weaned off by ≥ 8 weeks prior to Screening Visit 1
16. Subject with a history of bleeding diathesis or coagulopathy or subject who refuses blood transfusions
17. Subject working night shifts
18. Subject with a medical history of contraindications, anaphylactic reactions, or uncontrollable allergic reactions to contrast agents
19. Subject using active implantable medical devices (Implantable Cardioverter Defibrillator [ICD] or Cardiac Resynchronization Therapy Device [CRT-D], neuromodulation device, spinal cord stimulator, pressure reflector, etc.)
20. Subject with scheduled or planned surgery that may affect clinical investigation endpoints, in the opinion of the investigator
21. Subject has a documented condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement using the protocol-specified automatic/office blood pressure monitor (e.g., upper arm circumference outside cuff size ranges available by geography or arrhythmia that interferes with automatic monitor's pulse sensing and prohibits an accurate measurement).
22. Subject with documented confounding medical condition that may adversely affect the safety of the subject, in the opinion of the investigator (e.g. clinically significant peripheral vascular disease, aortic aneurysm, severe cardiac valve stenosis for which a significant reduction of blood pressure is contraindicated, or bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia,)
23. Subject with known unresolved history of drug use or alcohol dependency, lacks ability to comprehend or follow instructions, or would be unlikely or unable to comply with clinical investigation follow-up requirements
24. Subject currently enrolled in a concurrent investigational drug or device clinical investigation, unless approved by clinical investigation sponsor
25. 23)25) Pregnant, nursing, or planning to become pregnant during the course of the clinical investigation or follow-up. A negative pregnancy test is required for all women of child- bearing potential.
26. Subject who is unsuitable for the study for any reason as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in 24-h ambulatory systolic blood pressure | from baseline to 3 months post-procedure
  Change in 24-h ambulatory systolic blood pressure from baseline to 3 months post-procedure
Incidence of MAE within 3 months post-procedure | within 3 months post-procedure
  Incidence of MAE within 3 months post-procedure

SECONDARY OUTCOMES:
Changes in 24-h ambulatory systolic blood pressure | from baseline to 6, 12, and 24 months post-procedure
  Changes in 24-h ambulatory SBP from baseline to 6, 12, and 24 months post-procedure
Changes in 24-h ambulatory diastolic blood pressure | from baseline to 3, 6, 12, and 24 months post-procedure
  Changes in 24-h ambulatory DBP from baseline to 3, 6, 12, and 24 months post-procedure
Changes in office systolic blood pressure | from baseline to 1, 3, 6, 12, and 24 months post-procedure
  Changes in office SBP from baseline to 1, 3, 6, 12, and 24 months post-procedure
Changes in office diastolic blood pressure | from baseline to 1, 3, 6, 12, and 24 months post-procedure
  Changes in office DBP from baseline to 1, 3, 6, 12, and 24 months post-procedure
Incidence of achieving target office systolic blood pressure (< 140 mmHg) | from baseline to 1, 3, 6, 12, and 24 months post-procedure
  Incidence of achieving target office SBP (< 140 mmHg) from baseline to 1, 3, 6, 12, and 24 months post-procedure
Changes in heart rate | from baseline to 3, 6, 12, and 24 months post-procedure
  Changes in heart rate from baseline to 3, 6, 12, and 24 months post-procedure
Incidence of AEs, SAEs, ADE, and SADE | at 1, 3, 6, 12, and 24 months post-procedure
  Incidence of Adverse Events (AEs), SAEs, Adverse Device Effects (ADE), and Serious Adverse Device Effects (SADE) at 1, 3, 6, 12, and 24 months post-procedure
Incidence of MAE | at 6, 12, and 24 months post-procedure
  Incidence of MAEs at 6, 12, and 24 months post-procedure
Incidence of significant embolic event resulting in end-organ damage, incidence of renal artery perforation requiring intervention, incidence of renal artery dissection requiring intervention, incidence of vascular complications | at 1 month post-procedure
  Incidence of significant embolic event resulting in end-organ damage, incidence of renal artery perforation requiring intervention, incidence of renal artery dissection requiring intervention, incidence of vascular complications at 1 month post-procedure
Incidence of all-cause mortality | at 3, 6, 12, and 24 months post-procedure
  Incidence of all-cause mortality at 3, 6, 12, and 24 months post-procedure
Incidence of end-stage renal disease, incidence of ≥ 40% decline in eGFR, incidence of new myocardial infarction, incidence of new stroke, incidence of renal artery reintervention | at 1, 3, 6, 12, and 24 months post-procedure
  Incidence of end-stage renal disease, incidence of ≥ 40% decline in estimated glomerular filtration rate (eGFR), incidence of new myocardial infarction, incidence of new stroke, incidence of renal artery reintervention at 1, 3, 6, 12, and 24 months post-procedure
Incidence of major bleeding according to Thrombolysis in Myocardial Infarction (TIMI) definition | at 1, 3, 6, 12, and 24 months post-procedure
  Incidence of major bleeding according to Thrombolysis in Myocardial Infarction (TIMI) definition at 1, 3, 6, 12, and 24 months post-procedure (intracranial hemorrhage, ≥ 5 g/dL decrease in hemoglobin concentration, ≥ 15% absolute decrease in hematocrit, or death due to bleeding within 7 days of procedure)
Incidence or increase in serum creatinine > 50% | at 1, 3, 6, 12, and 24 months post-procedure
  Incidence or increase in serum creatinine > 50% at 1, 3, 6, 12, and 24 months post-procedure
Incidence of new renal artery stenosis > 70% | at 3 months post-procedure
  Incidence of new renal artery stenosis > 70% at 3 months post-procedure, as assessed by Computed Tomography (CT), Magnetic Resonance Angiography (MRA), or Doppler Ultrasonography (DUS)
Incidence of hospitalization for hypertensive crisis not related to confirmed non-adherence or the CIP | at 1, 3, 6, 12, and 24 months post-procedure
  Incidence of hospitalization for hypertensive crisis not related to confirmed non-adherence or the CIP at 1, 3, 6, 12, and 24 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tsioufis, Professor, Principal Investigator — National and Kapodistrian University of Athens, Greece; Felix Mahfoud, Professor, Study Director — Saarland University Hospital, Homburg; Massimo Volpe, Professor, Study Director — University of Roma La Sapienza; Jacek Kadziela, Professor, Principal Investigator — Narodowy Instytut Kardiologii Stefana kardynała Wyszyńskiego, Poland
Locations (1):
- University of Athens Hippocratio Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No